CLINICAL TRIAL: NCT06144008
Title: ESCAPE (Evaluating Surge Capacity And PrEparedness): a Multicenter Study on Recruiting Students as Surge Capacity Workforce in the Event of a Pandemic
Brief Title: ESCAPE (Evaluating Surge Capacity And PrEparedness)
Acronym: ESCAPE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. B. Zwissler, Head of the Department of Anaesthesiology of the University Hospital of Munich, Ludwig-Maximilians - University of Munich
Other Study IDs: Klinikum Großhadern
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Disaster Medicine; Delivery of Health Care
Keywords: Surge capacity; Disaster medicine; pandemic preparedness; Hospital volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical experts in departments at risk: Expert healthcare workers at the Munich University Hospital within departments potentially affected by a major medical incident that could benefit from student surge capacity workforce. The following departments are included: Emergency Department, Intensive Care Units, Intermediate Care Units, Medical and Surgical wards, Department for Microbiology, Department for Infectious Diseases, Department for Laboratory Medicine, Antibiotic Stewardship Team, Department for Tropical Medicine, Max-von-Pettenkofer Institute, Institute for Emergency Medicine, Faculty Dean's office.
  Interventions: Behavioral: Answering questionnaire
- Students: Medical students from all medical faculties in Germany to be questioned on their willingness to partake in clinical work as surge capacity work force in the context of a potential major medical incident.
  Interventions: Behavioral: Answering questionnaire

INTERVENTIONS:
Behavioral: Answering questionnaire — A questionnaires for each group has been developped and will be distributed for voluntary and anonymous completion.

SUMMARY:
The ESCAPE study intends to assess the possibility of recruiting students as surge capacity work force in hospitals in the event of a major medical incident such as an epidemic or pandemic.

DETAILED DESCRIPTION:
The ESCAPE study intends to assess the possibility of recruiting students as surge capacity work force in hospitals in event of a major medical incident such as an epidemic or pandemic. The study consists of two parts:

* To identify the need for student surge capacity work force in relevant departments most affected by major medical incidents (e.g. Emergency Department, Intensive Care Unit, etc.). This part also raises the question of which tasks can be delegated to such a surge capacity workforce and which training may be required to prepare for such tasks.
* To identify and quantify the willingness of students to enroll as surge capacity workforce, identifying which tasks they would be willing to perform and which organisational framework is required for their work (training, insurance, pay, etc.).

Both subparts as planned as questionnaires to be completed voluntarily and anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Medical experts (heads of departements and other management positions) working in selected departments that are typically affected by major medical incidents at the time of questionnaire roll-out.
* Medical students >18 years of age of any year enrolled in the year 2023-2024 in any of the 38 medical faculties in Germany

Exclusion Criteria:

* none, as questionnaire participation was achieved by invitation of eligible volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Heads of departments typically affected by major medical incidents. These include: Emergency Department, Intensive Care Units, Intermediate Care Units, Medical and Surgical wards, Department for Microbiology, Department for Infectious Diseases, Department for Laboratory Medicine, Antibiotic Stewardship Team, Department for Tropical Medicine, Max-von-Pettenkofer Institute, Institute for Emergency Medicine, Faculty Dean's office. Included were: heads of departments and other members of leadership from the medical staff, nursing staff and other supporting staff.
  * Medical students (aged 18 and over) in any year, currently studying at any of the 38 medical faculties in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Student surge capacity workforce needed | baseline
  Is the general opinion that a student workforce would be beneficial in the context of a major medical incident?

SECONDARY OUTCOMES:
Student willingness to work as student surge capacity workforce | baseline
  Are medical students willing to be involved as surge capacity workforce?
Tasks to be delegated to surge capacity workforce | baseline
  What tasks can be delegated to a student workforce and what training is required to safely delegate these?
Organisational framework in which to embed surge capacity workforce | baseline
  What organisational aspects need to be addressed in setting up a student surge capacity workforce?

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Zwissler, Prof, MD, Principal Investigator — Ludwigs-Maximilians-University Munich; Martin Fischer, Prof, MD, Principal Investigator — Ludwigs-Maximilians-University Munich
Locations (1):
- Department of Anaesthesiology of the University Hospital of Munich, Munich, Germany